CLINICAL TRIAL: NCT00002057
Title: Nystatin Pastilles for the Prevention of Oral Candidiasis in Patients With AIDS or ARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: 026A; 4
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: Candidiasis, Oral; HIV Infections
Keywords: Nystatin; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Candidiasis, Oral
MeSH Terms: conditions — Candidiasis, Oral; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Nystatin

INTERVENTIONS:
Drug: Nystatin

SUMMARY:
To determine a safe, effective, and convenient dosing schedule for nystatin pastilles in the prevention of oral candidiasis in patients with AIDS or AIDS related complex (ARC) (group III or IV, CDC classification).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Systemic or oral antibiotics.
* Experimental drugs (IND drugs) which are targeted specifically against the AIDS (group IV CDC classification) virus or stimulate the immune system.

Patients with the following conditions are included:

* AIDS or AIDS related complex (ARC) (HIV infection Group 3 or 4, CDC classification) who have had culture-proven oral candidiasis clinically cured within 7 days of study entry and are likely to be compliant for the 20 weeks of nystatin pastille prophylaxis.
* Able to follow instructions regarding the use of a pastille.
* Patients entering part II of this study (randomized double-blind) must have been clinically cured of oral candidiasis within 1 - 7 days of entry into this randomized study.
* Oral lesions such as Kaposi's sarcoma, herpes zoster, and herpes simplex can be enrolled.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Systemic candidiasis.
* Hypersensitivity to nystatin.
* Suspected or proven candidal esophagitis.

Patients with the following are excluded:

* Systemic candidiasis.
* Projected survival of less than 6 months.
* Unable to maintain a pastille in the buccal cavity for approximately 20 minutes twice a day.
* Hypersensitivity to nystatin.
* Suspected or proven candidal esophagitis.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Birmingham Veterans Administration Med Ctr / Univ of Alabama, Birmingham, Alabama
  - Bristol - Myers Squibb Co, Princeton, New Jersey